CLINICAL TRIAL: NCT00091546
Title: Genetic and Environmental Pathogenesis of PPH
Brief Title: Genetic and Environmental Characteristics of Primary Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jim Loyd, Professor, Vanderbilt University
Other Study IDs: 166; P01HL072058 (NIH)
Record Dates: First submitted 2004-09-10; First posted 2004-09-13 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Lung Diseases; Hypertension, Pulmonary
MeSH Terms: conditions — Lung Diseases; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Specimens from 100 families affected by PPH
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to identify the modifying genes and environmental features that regulate the clinical expression of mutations in bone morphogenetic protein receptor 2 (BMPR2); to develop the understanding of how BMPR2 mutations result in disease; and to identify the undiscovered genetic mutations that cause primary pulmonary hypertension (PPH).

DETAILED DESCRIPTION:
BACKGROUND:

PPH is a progressive disease that causes obstruction of the smallest arteries in the lungs, which often leads to heart failure. It threatens the lives of thousands of individuals. PPH affects both genders at any age, although females are affected twice as often as males. In a recent important advance, mutations in BMPR2 were associated with both familial and sporadic PPH. Because only 20% of people with a BMPR2 mutation ever develop PPH, other genes or modifying biologic events must contribute to the clinical development of the disease. PPH was recently renamed Idiopathic Pulmonary Arterial Hypertension or Familial Pulmonary Arterial Hypertension.

DESIGN NARRATIVE:

This study will utilize a database and specimen bank developed from 100 families affected by PPH across the United States. In families with genetic mutations not yet identified, changes in the BMPR2 gene will be studied, including in the promoter and intronic regions, and chance recombination events that could confirm another locus near 2q33 will be examined. New methods will look for modifier genes in large families with known mutations; examine kindreds for mitochondrial DNA haplotypes; and test candidate genes, including NOS-1, NOS-3, and the serotonin transporter. This study will determine the functional mechanisms by which variations found in the BMPR2 alleles alter BMP signal transduction by defining the biochemical effects of the mutant proteins on signaling pathways. In addition, the study will examine the perceived risks and benefits of clinical genetic testing and counseling in individuals from families at high risk for PPH and will determine how this new information might be most helpful to these individuals and their families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPH, or family members of individuals diagnosed with PPH, for inclusion in the database and specimen bank

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Database and specimen bank developed from 100 families affected by PPH
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2003-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
New development of pulmonary arterial hypertension (penetrance), age of onset, and survival | Measured through genetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: James Loyd, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cogan JD, Vnencak-Jones CL, Phillips JA 3rd, Lane KB, Wheeler LA, Robbins IM, Garrison G, Hedges LK, Loyd JE. Gross BMPR2 gene rearrangements constitute a new cause for primary pulmonary hypertension. Genet Med. 2005 Mar;7(3):169-74. doi: 10.1097/01.gim.0000156525.09595.e9. PMID 15775752
- [Background] Meyrick BO, Friedman DB, Billheimer DD, Cogan JD, Prince MA, Phillips JA 3rd, Loyd JE. Proteomics of transformed lymphocytes from a family with familial pulmonary arterial hypertension. Am J Respir Crit Care Med. 2008 Jan 1;177(1):99-107. doi: 10.1164/rccm.200703-499OC. Epub 2007 Oct 11. PMID 17932379
- [Background] Phillips JA 3rd, Poling JS, Phillips CA, Stanton KC, Austin ED, Cogan JD, Wheeler L, Yu C, Newman JH, Dietz HC, Loyd JE. Synergistic heterozygosity for TGFbeta1 SNPs and BMPR2 mutations modulates the age at diagnosis and penetrance of familial pulmonary arterial hypertension. Genet Med. 2008 May;10(5):359-65. doi: 10.1097/GIM.0b013e318172dcdf. PMID 18496036
- [Background] Newman JH, Phillips JA 3rd, Loyd JE. Narrative review: the enigma of pulmonary arterial hypertension: new insights from genetic studies. Ann Intern Med. 2008 Feb 19;148(4):278-83. doi: 10.7326/0003-4819-148-4-200802190-00006. PMID 18283205
- [Result] Cogan JD, Pauciulo MW, Batchman AP, Prince MA, Robbins IM, Hedges LK, Stanton KC, Wheeler LA, Phillips JA 3rd, Loyd JE, Nichols WC. High frequency of BMPR2 exonic deletions/duplications in familial pulmonary arterial hypertension. Am J Respir Crit Care Med. 2006 Sep 1;174(5):590-8. doi: 10.1164/rccm.200602-165OC. Epub 2006 May 25. PMID 16728714
- [Derived] Johnson JA, Vnencak-Jones CL, Cogan JD, Loyd JE, West J. Copy-number variation in BMPR2 is not associated with the pathogenesis of pulmonary arterial hypertension. BMC Med Genet. 2009 Jun 16;10:58. doi: 10.1186/1471-2350-10-58. PMID 19531247